CLINICAL TRIAL: NCT06856486
Title: Sulforaphane-Smart® on Lipid and Glucose Metabolism, Inflammation, Adiposity and Microbiome of Overweight Adults "SANO"
Brief Title: Acute Intervention with Sulforaphane-Smart®
Acronym: SANO-Acute
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mª Jesús Periago (Other)
Collaborators: Ingredalia Company (Unknown); Spanish National Research Council (CEBAS-CSIC) (Unknown)
Responsible Party: Sponsor-Investigator, Mª Jesús Periago, PhD Full Professor of Food Science and Nutrition, Universidad de Murcia
Organization: Universidad de Murcia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SANO Bioavailability Project; CPP2022-009528 (Other: Ministerio de Ciencia, Innovación y Universidades)
Record Dates: First submitted 2025-02-10; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Glucosinolates; Isothiocyanates; Sulforaphane; bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sulforaphan-Smart® formula (Experimental): Intake of the Sulforaphan-Smart® formula to evaluate its pharmacokinetics in biological samples of plasma and urine.
  Interventions: Dietary Supplement: Sulforaphan Smart®

INTERVENTIONS:
Dietary Supplement: Sulforaphan Smart® — Fasting volunteers will intake the Sulforaphan Smart® pill, and blood and urine samples will be taken at the beginning of the intervention (Time 0 hours, before intake the pill), and 6 and 24 hours after its intake the pills (Time 6 hours and Time 24 hours) to measure the biomarkers related to the bioavailability of GSL/ITCs.

SUMMARY:
The Sulforaphane-Smartt® formula is a pill, patented by the company INGREDALIA, prepared with broccoli by-products which have been concentrated and enriched in glucosinolates/isothiocyanates (GLS/ITCs).

The goal of this intervention study with the Sulforaphane-Smartt® formula is to study the bioavailability of the bioactive compounds in normal weight and overweight adults. The main questions it aims to answer are:

* Determine the absorption curve of the bioactive compounds (GLS/ITCs).
* Analyze the metabolites in plasma and urine of the GLS/ITCs to know the bioavailability.

This acute intervention is designed to take a single fasting dose of Sulforaphan-Smart®, collecting plasma and urine samples to study free and conjugated metabolites of GLS/ITC.

There is not a comparison group, since the acute intervention study with the Sulforaphane-Smart® is designed to determine the bioavailability of the bioactive compounds (GLS/ITCs).

DETAILED DESCRIPTION:
Sulforaphan-Smart® is a formula patented by the company INGREDALA (patented by INGREDALIA: EP3123874B1). This clinical trial will provide information about the bioavailability of the bioactive compounds of this formula (GLS/ITCs). The results of this research project will give us the possibility of obtaining a nutraceutical product based on the increasing the technology readiness level (TRL) from the current TRL5 to TRL6-7.

An acute intervention study will be conducted with 20 participants, normal-weight and overweight volunteers of both sexes, to evaluate the bioavailability and the absorption curve of the GSL/ITCs by the analysis of metabolites in urine and blood. These metabolites are considered biomarkers of intake and will allow to study the bioavailability of the bioactive compounds of the Sulforaphan-Smart® formula.

Participants will be informed about the study design and activities and will signed the informed consent. They will follow a diet free of Cruciferous during 72 h before the beginning of the study, as washout period. After that participants will take a single dose of Sulforaphane-Smart® pill on a fasting regimen. To evaluate the bioavailability of the bioactive compounds (GLS/ITCs) blood samples will be withdrawn at 0, 6 and 24 h, whereas urine samples will be collected at 0, 6 and 24 h after ingestion of Sulforaphan-Smart® pill.

Free and conjugated metabolites will be analysed in plasma and urine by UHPLC-QqQ-MS/MS following their fragmentation patterns, with the aim to evaluate the bioavailability of the GSL/ITCs of the Sulforaphan-Smart® formula.

ELIGIBILITY:
Inclusion Criteria:

* BMI: normal weight or overweight volunteers
* No digestive or intestinal diseases
* Age between 20 and 45 years old
* Not having antibiotics during the previous three months
* Not having pharmacological treatment
* Not being smokers
* Not following restrictive diets (vegetarian/vegan diet) or nutritional supplement

Exclusion Criteria:

* BMI: low weight and obesity
* Age different from that required
* Digestive or intestinal diseases
* Having antibiotics during the previous three months
* Having pharmacological treatments
* Following restrictive diets (vegetarian/vegan diet) or nutritional supplement
* Smoker
* Menopause

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Characterization of free and conjugated metabolites of GLs/ITCs in urine and plasma at the beginning of the intervention (Time 0 hours) | Analysis of metabolites of GSL/ITCs before intake the Sulforaphane-Smart pill.
  Samples of blood and urine will be taken before the intake of the pill. The investigators will analyse the profile of free and conjugated metabolites in plasma and urinary using UHPLC-QqQ-MS/MS following their fragmentation patterns.
Characterization of free and conjugated metabolites of GLs/ITCs in urine and plasma after 6 hours of the intake of pill (Time 6 hours) | Analysis of metabolites of GSL/ITCs after 6 hours taking the Sulforaphane-Smart pill.
  Samples of blood and urine will be collected after 6 hours taking the pill. The investigators will analyze metabolites in plasma and urinary using UHPLC-QqQ-MS/MS following their fragmentation patterns.
Characterization of free and conjugated metabolites of GLs/ITCs in urine and plasma after 24 hours of the intake of pill (Time 24 hours) | Analysis of metabolites of GSL/ITCs after 24 hours taking the Sulforaphane-Smart pill.
  Samples of blood and urine will be taken 24 hours after taking the pill. The investigators will analyse the profile of free and conjugated metabolites in plasma and urinary using UHPLC-QqQ-MS/MS following their fragmentation patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Rocío González Barrio, Principal Investigator — Universidad de Murcia; María Jesús Periago Castón, Principal Investigator — Universidad de Murcia
Locations (1):
- Edificio Pleyades-Vitalys 5ª y 6ª planta, Campus Universitario, Espinardo, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Review about the clinical trials with broccoli sprouts or sulforaphane to investigate the beneficial effect for human health — https://doi.org/10.3389/fnut.2021.648788